CLINICAL TRIAL: NCT05739617
Title: Combining Sonography to Explore the Therapeutic Effect and Mechanism of a Comprehensive Respiratory Training Exercise Program on Cardiorespiratory Endurance and Airway Muscle Function in Obstructive Sleep Apnea
Brief Title: Comprehensive Respiratory Training Exercise Program in Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-111-079
Record Dates: First submitted 2023-02-08; First posted 2023-02-22 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Hygiene Education (Sham Comparator): Participants will received once per month of sleep hygiene education for three months.
  Interventions: Other: Sleep hygiene education
- Comprehensive Respiratory Training Exercise Program (Experimental): Participants will received Comprehensive Respiratory Training Exercise Program twice per weeks for three months.
  Interventions: Other: Comprehensive Respiratory Training Exercise Program

INTERVENTIONS:
Other: Comprehensive Respiratory Training Exercise Program — This comprehensive respiratory training exercise program consists of four main components, including oropharyngeal muscle training, respiratory muscle training, aerobic exercise, and sleep hygiene education.
  Arms: Comprehensive Respiratory Training Exercise Program
Other: Sleep hygiene education — Sleep hygiene education
  Arms: Sleep Hygiene Education

SUMMARY:
Obstructive sleep apnea (OSA) is a multi-factorial sleep disorder. Complete collapse or partial collapse in the airway increases the risk of developing cardiovascular and kidney-related disease in OSA patients. Resulting in an increase in medical expenses and workload for the healthcare worker. Multilevel of upper airway muscles especially the genioglossus muscle showed to contribute to airway obstruction as it fatigues easily. The endurance level of OSA patients was shown to be significantly lower. Therefore, the goal of this experimental study is to assess the feasibility and effectiveness of a comprehensive respiratory training exercise program on cardiorespiratory endurance, airway muscle function, and sleep parameters in patients with obstructive sleep apnea (OSA). Aside from exploring the therapeutic effect, the results of the study will be used to explore the mechanism of the treatment in relation to the changes in the OSA severity.

DETAILED DESCRIPTION:
Newly diagnosed OSA subjects, aged 20-65 years old, and with body mass index between 18-30 kg.m-2 will be recruited. The participants will be randomly divided into the control group (sleep hygiene education) and the intervention group (comprehensive respiratory training exercise program). Participants from the intervention group will undergo 3 months of a comprehensive respiratory training exercise program while the control group will be provided sleep hygiene education. Polysomnography (PSG), cardiopulmonary exercise testing, sonography (during the awake stage, functional tasks, Müller's maneuver, and natural sleep), tongue strength and tongue endurance assessment, jaw strength measurement, Computed Tomography (CT), Drug-Induced Sleep Endoscopy (DISE), respiratory muscle strength, pulmonary function test, and sleep quality questionnaires will be collected before and after 3 months of intervention.

Expected contribution to clinical medicine

* The feasibility of this comprehensive respiratory training exercise program in improving cardiorespiratory endurance, leading to an increase in the survival rate and reduced risk of cardiovascular disease of OSA patients.
* Based on the ultrasound's findings in the awake stage (normal breathing, functional tasks, and Müller's maneuver) and overnight sleep, allow a better understanding of the effects of these exercises on the changes of tongue and oropharyngeal structures during the static and dynamic stages.
* The practicability of the ultrasound assessment in the clinical setting on OSA patients is to identify the changes in the tongue and oropharyngeal structures. Based on ultrasound image capture, it provides individualized and precise training by modifying the training and providing feedback to OSA patients during their exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with OSA (AHI≥ 5 events per hour)
* Age between 20 to 65 years old
* BMI of 18-30 kg.m-2

Exclusion Criteria: Diagnosed with any of the following diseases below:

* Central or mixed types of sleep apnea
* Neuromuscular disease
* Severe cardiovascular disease
* Active psychiatric disease
* Head or neck disease or cancer
* Structural abnormalities over the upper respiratory airway
* Performed any operation or treatment over the neck before
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea-Hypopnea Index (AHI) | Baseline to 3 months (post-training)
  The apnea-hypopnea index will be obtained from the overnight Polysomnography (PSG) study. PSG will be performed in the sleep center of National Cheng Kung University Hospital. Less than 5 events/hour indicates normal; AHI between 5-14 events/hour indicates mild Obstructive Sleep Apnea(OSA); AHI between 15-30 events/hour indicates moderate OSA; and AHI more than 30 events/hour indicates severe OSA.
Change in Oxygen Desaturation Index (ODI) | Baseline to 3 months (post-training)
  The average number of desaturation episodes per hour (oxygen desaturation index) will be obtained from the overnight Polysomnography (PSG) study. A decrease in the mean oxygen saturation of ≥4% that lasts for at least 10 seconds indicates an episode of desaturation.
Change in Maximum Oxygen Consumption (Vo2max) | Baseline to 3 months (post-training)
  Maximum oxygen consumption (Vo2max) will be measured using Cardiopulmonary Exercise Testing (CPET) which will be performed on a static bicycle. The average value of Vo2max in adults is approximately 27-48 mL/kg/min. A greater Vo2max value indicates a better physical fitness level.
Change in Tongue Muscle Thickness | Baseline to 3 months (post-training)
  Sonography will be performed over the participant's neck region to assess the changes in tongue muscle thickness during normal breathing, Müller's maneuver, functional tasks, and natural sleep.
  The data on tongue thickness will be presented in millimeters. A greater value indicates a thicker in tongue.
Change in Tongue Muscle Stiffness | Baseline to 3 months (post-training)
  Ultrasound shear-wave elastography will be performed to assess the changes in tongue-based stiffness. The data will be presented in kPa, with a greater value indicating an increase in tongue stiffness. The minimum value is 0 kPa and the maximum value is 220 kPa.
Change in Tongue Muscle Strength | Baseline to 3 months (post-training)
  The tongue muscle strength will be measured using an Iowa Oral Performance Instrument (IOPI) device, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA). The minimum score is 0 and a higher score indicates stronger in tongue muscle strength.
Change in Tongue Muscle Endurance | Baseline to 3 months (post-training)
  The tongue muscle endurance will be measured using an Iowa Oral Performance Instrument (IOPI) device, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA). The data will be presented in seconds. The longer the duration of holding (more than 10 seconds), the greater in the tongue muscle endurance.
Change in Jaw strength | Baseline to 3 months (post-training)
  Jaw strength will be measured using a 'handheld' dynamometer (MicroFET○R2, Hoggan Scientific, USA). The data will be presented in kilogram-weight. The minimum score is 0 and a higher score indicates stronger in jaw strength.
Change in Pharyngeal Airway Volume | Baseline to 3 months (post-training)
  Computer Tomography (CT) will be performed. The pharyngeal airway volume will be calculated from the hard palate to the epiglottis and the data will be presented in cm3. The minimum score is 0 and a higher score indicates greater in pharyngeal airway volume.
Change in Cross Section Area on the Tip of Epiglottis | Baseline to 3 months (post-training)
  Computer Tomography (CT) will be performed. Cross section area on the tip of the epiglottis was measured and the data will be presented in cm2. The minimum score is 0 and a higher score indicates greater in the cross-sectional area of the region.
Change in Anterior to Posterior Distance on the Tip of the Epiglottis | Baseline to 3 months (post-training)
  The distance between the anterior and posterior pharyngeal wall on the tip of the epiglottis will be measured and presented in cm. The minimal value will be 0 and the greater value indicates a greater distance between the anterior to posterior in this area.
Change in Lateral Distance on the Tip of Epiglottis | Baseline to 3 months (post-training)
  The distance between the lateral distance on the tip of the epiglottis will be measured and presented in cm. The minimal value will be 0 and the greater value indicates a greater distance between the lateral wall.
Change in daytime sleepiness | Baseline to 3 months (post-training)
  Epworth Sleepiness Score(ESS) will be used to measure the daytime sleepiness of OSA patients. The total score of ESS range from 0-24. A score greater than 10 indicates greater daytime sleepiness.
Change in Drug-induced Sleep Endoscopy (DISE) | Baseline to 3 months (post-training)
  The level of obstruction, the degree of obstruction, and the configuration of the obstructive will be identified through the drug-induced sleep endoscopy. The degree of obstruction ranged from 0 to 2. 0: no obstruction; 1: partial obstruction; 2: complete obstruction.
Change in sleep quality | Baseline to 3 months (post-training)
  Sleep quality will be measured using Pittsburgh Sleep Quality Index (PSQI).The total score ranges from 0 to 21 with a higher total score equal to or more than 5 indicating worse sleep quality.

SECONDARY OUTCOMES:
Change in Maximal Inspiratory Pressure (PImax) | Baseline to 3 months (post-training)
  For respiratory muscle strength, maximal inspiratory pressure (PImax) will be measured using Respiratory Pressure Meter. Data will be presented in cmH2O. The minimal score will be 0, and a higher value indicates stronger in the inspiratory muscle.
Change in Maximal Expiratory Pressure (PEmax) | Baseline to 3 months (post-training)
  For respiratory muscle strength, maximal expiratory pressure (PEmax) will be measured using Respiratory Pressure Meter. Data will be presented in cmH2O. The minimal score will be 0, and a higher value indicates stronger in the expiratory muscle.
Change in forced vital capacity (FVC) % predicted | Baseline to 3 months (post-training)
  The respiratory muscle function on the forced vital capacity (FVC) % predicted will be collected using spirometry. The normal value is between 80% to 120%; mild abnormality: is 70-79%; moderate abnormality: is 60-69%; severe abnormality: is less than 60%.
Change in Forced Expiratory Volume in one second (FEV1)/ forced vital capacity(FVC) % | Baseline to 3 months (post-training)
  The respiratory muscle function on the Forced Expiratory Volume in one second (FEV1)/ forced vital capacity(FVC) will be collected using spirometry. The normal value for the FEV1/FVC % is equal to or greater than 70%; mild abnormality: 60-69%; moderate abnormality: 50-59%; severe abnormality: less than 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No